CLINICAL TRIAL: NCT05112263
Title: Tofacitinib Versus Cyclosporine for Steroid Refractory Acute Severe Ulcerative Colitis: An Open Label Randomized Study
Brief Title: Tofacitinib Versus Cyclosporine for Steroid Refractory Acute Severe Ulcerative Colitis
Acronym: TOCASU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vishal Sharma, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/2021/000641
Record Dates: First submitted 2021-10-26; First posted 2021-11-08 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: Intravenous Cyclosporine 2 mg/kg continuous infusion for 5-7 days and then shifted to oral cyclosporine 4 mg/kg/day in two divided doses for 12 weeks
  Interventions: Drug: Cyclosporine
- Group B (Experimental): Oral Tofacitinib 10 mg TDS for 3 days, and then 10 mg BD to complete 8 weeks followed by 5 mg BD till follow-up (14 weeks)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — For the tofacitinib the dose of 10 mg BD will be administered for 8 weeks (10 mg TDS for initial three days) and then reduced to 5 mg BD for the period of study
  Arms: Group B
Drug: Cyclosporine — : Intravenous Cyclosporine 2 mg/kg continuous infusion for 5-7 days and then shifted to oral cyclosporine 4 mg/kg/day in two divided doses for 12 weeks.Those who respond with intravenous cyclosporine will be shifted to oral cyclosporine 4 mg/kg for 12 weeks while the thiopurine dose is adjusted to the patient's weight
  Arms: Group A

SUMMARY:
This randomised trial plans to compare oral tofacitinib with intravenous cyclosporine in patients with acute severe ulcerative colitis who have failed to respond to intravenous steroids

ELIGIBILITY:
Inclusion Criteria:

Patients admitted with Acute severe ulcerative colitis as defined by Modified Truelove and Witts Criteria WITH Failure to respond to intravenous steroids (Hydrocortisone 100 mg IV QID OR IV Methylprednisolone 60 mg IV OD) as defined by

* Day 3 non-response as per Oxford criteria (stool frequency of > 8/day, OR stool frequency between 3-8 with CRP > 45 mg/L PLUS
* Ongoing activity as defined by Partial Mayo Score of > 3 (rectal bleeding sub-score of >1)
* Decision to start second line therapy (within 5-7 days of starting intravenous steroids)

Exclusion Criteria:

* Age <18, Age > 65 years

  * E1 disease (involvement distal to rectosigmoid junction only)
  * Crohn's disease
  * Contraindication to intravenous cyclosporine or oral tofacitinib

    * Renal failure, uncontrolled hypertension, seizure disorder,and uncorrected hypomagnesemia (<1.5 mg/L)
    * Previous thrombosis, or prothrombotic state, on oral contraceptive, history of herpes zoster, active TB, active hepatitis, past opportunistic infections, h/o diverticulitis, Age >50 plus at least one cardiac risk factor
  * Patient wants treatment with intravenous infliximab or wants surgery
  * Underlying sepsis or active infection (Enteric infections, Clostridium difficile, active hepatitis B or C, Tuberculosis, zoster, CMV disease)
  * Toxic megacolon, previous dysplasia or any indication of immediate surgery
  * Known malignancy
  * Pregnancy or Lactation
  * Unwilling to provide consent or for follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 14 weeks
  I) At Day 7 Absence of clinical response at day 7 (as defined by Partial Mayo of > 3)
  II) By Day 98
  1. Relapse (Partial Mayo Score of 3 or more) between day 7 and day 98 requiring additional therapy
  2. Absence of steroid free remission at 14 weeks (Mayo < 2 with MES 1 or less)
  3. Need for colectomy, third line medical rescue or biologics or mortality
  4. Serious adverse effect needing interruption of treatment

SECONDARY OUTCOMES:
Clinical response | 7 days
  Partial Mayo <4
Absence of steroid free remission | day 98
  Mayo score of more than 2 with endoscopic sub-score of more than 1
Colectomy free survival | 98 days
  No need for colectomy
Time to clinical response | 98 days
  Partial Mayo of 3 or less
Endoscopic healing | Day 98
  Mayo endoscopic sub-score of 1 or less
Serious adverse effects | 98 days
  requiring hospitalization, cessation of treatment and events like cardiovascular events, pulmonary embolism, venous thrombosis, any infection, malignancy, gastrointestinal perforation

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Sharma, Principal Investigator — PGIMER Chandigarh; Vineet Ahuja, Principal Investigator — AIIMS Delhi

IPD SHARING:
Plan to Share IPD: No
The anonymised participant data may be shared on reasonable request